CLINICAL TRIAL: NCT03648294
Title: Long-term Blood Pressure Outcome After Unilateral Adrenalectomy for Primary Hyperaldosteronism
Acronym: Hyperaldo
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0040
Record Dates: First submitted 2018-08-21; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Adrenalectomy; Status
Keywords: blood pressure
MeSH Terms: interventions — Adrenalectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: adrenalectomy for primary addosteronism — All of the clinical and biological data were retrospectively compiled from the patient computerized record. The variables analyzed were: age, sex, body mass index (BMI), PAH discovery circumstances, pre- and postoperative systolic and diastolic blood pressure assessments, number of pre-hypertensive antihypertensive drug - and postoperatively, the laterality, the size and nature of the lesions, the operating time, the surgical technique used. The biological data evaluated were pre- and postoperative plasma and plasma creatinine, preoperative serum aldosterone concentrations, plasma renin activity, and preoperative aldosterone / renin ratio. Hypokalemia was defined as serum concentration below 3.5 mmol / L.

SUMMARY:
To evaluate long-term results of adrenalectomy for primary aldosteronism (PA) and to identify prognostic factors associated.

Exhaustive retrospective review of all consecutive patients undergoing adrenalectomy for PA between 2002 and 2013 in our department. All patients underwent preoperative: clinical evaluation (age, sex, height, weight, systolic and diastolic BP under treatment, identification of anti-hypertension treatment), biological evaluation (potassium, renin, aldosterone) and radiological evaluation (CT and/or MRI). Blood pressure was assessed postoperatively at 1 month, 1 year, then at the date of the latest news. The patients were classified into three categories: cured (no antihypertensive therapy in postoperative associated with strictly lower blood pressures of 140/90mmHg), improved (decreased number of drugs or number unchanged but with better blood pressure control), and refractory (no change in the number of drug and blood pressure, or deterioration of one or other of these two parameters).

DETAILED DESCRIPTION:
To evaluate long-term results of adrenalectomy for primary aldosteronism (PA) and to identify prognostic factors associated.Exhaustive retrospective review of all consecutive patients undergoing adrenalectomy for PA between 2002 and 2013 in our department. All patients underwent preoperative: clinical evaluation (age, sex, height, weight, systolic and diastolic BP under treatment, identification of anti-hypertension treatment), biological evaluation (potassium, renin, aldosterone) and radiological evaluation (CT and/or MRI). Blood pressure was assessed postoperatively at 1 month, 1 year, then at the date of the latest news. The patients were classified into three categories: cured (no antihypertensive therapy in postoperative associated with strictly lower blood pressures of 140/90mmHg), improved (decreased number of drugs or number unchanged but with better blood pressure control), and refractory (no change in the number of drug and blood pressure, or deterioration of one or other of these two parameters).

ELIGIBILITY:
Inclusion Criteria:

* Patients >25 years and <80 years patients undergoing adrenalectomy for PA
* All patients underwent preoperative: clinical evaluation (age, sex, height, weight, systolic and diastolic BP under treatment, identification of anti-hypertension treatment), biological evaluation (potassium, renin, aldosterone) and radiological evaluation (CT and/or MRI).

Exclusion Criteria:

* patients <25 years
* patients > 80 years

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between 2002 and 2013, the investigators evaluated all patients receiving adrenalectomy and extracted data on PAH patients. The diagnosis was made on the presence of hypertension (all stages combined), an autonomous hyperproduction of aldosterone and sometimes hypokalemia (n = 32). HTA was defined, in accordance with the recommendations of the Haute Autorité de Santé and the French Society of Arterial Hypertension (blood pressure greater than or equal to 140/90 mmHg)
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Adrenalectomy for primary hyperaldosteronism | 1 year
  The objective of this study is to evaluate the course of the disease associated with long-term outcomes of adrenalectomy for the treatment of PAH, with a retrospective analysis of patient data!

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Saint, MD, PhD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No